CLINICAL TRIAL: NCT02406391
Title: Adherence to Screening and Follow-up Diagnostic and Treatment Services for Cervical Cancer Prevention
Brief Title: Adherence to Preventive Care for Cervical Cancer
Acronym: Adh-NYC-EP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brookdale University Hospital Medical Center (Other)
Responsible Party: Principal Investigator, Michele Follen, Chair of Department of Obstetrics and Gynecology, Brookdale University Hospital Medical Center
Other Study IDs: 14-40
Record Dates: First submitted 2015-03-16; First posted 2015-04-02 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Cancer; Cervical Precancer; Adherence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
In the United States, the highest incidence of cervical cancer occurs in inner city urban centers, rural areas, the deep South, Appalachia and the U.S.-Mexico border. The goal of this study is to study predictors of adherence among patients seeking care at an inner city medical center in New York City and the U.S. Mexico border for cervical cancer prevention, namely, Pap smears and colposcopy exams.

DETAILED DESCRIPTION:
Because there are multiple pathways through which a person is influenced to seek and receive care, the investigators will conduct interviews with patients seeking care for cervical cancer prevention at an inner city medical center. The investigators will ask questions related to previous screening, diagnostic, and treatment practices as well as barriers experienced in seeking such care. The investigators will also explore patients' level of resiliency and coping as predictors of adherence to timely care. Furthermore, among immigrants, questions about acculturation and discrimination will be asked. Additional measures of socioeconomic status, such as education, income and occupation will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* women who are at least 21 years old
* are seeking care for a Pap smear exam
* are seeking care for a colposcopy exam for the first time
* are not pregnant by self-report
* are able to provide informed consent

Exclusion Criteria:

* women who do not meet the above eligibility criteria
* women who have no prior history of a hysterectomy
* women who have previously participated in this study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients who present to the gynecology clinic for a Pap smear exam or a colposcopy exam following an abnormal Pap smear.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to screening, colposcopy and follow-up treatment | 1-2 hour interview during clinic visit and review of patients' medical records during surveillance period (up to 2 years)
  A survey will be administered to patients who present for a routine Pap smear exam, a follow-up colposcopy exam. Medical records will be reviewed to document adherence to treatments post-colposcopy

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Principal Investigator — Brookdale University Hospital and Medical Center
Locations (3):
- United States (3):
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - University of Texas at El Paso, El Paso, Texas
  - Texas Tech University Health Science Center, El Paso, Texas